CLINICAL TRIAL: NCT01355601
Title: Effect of Carbohydrates From Nutritional Beverages in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to slow recruitment. 41 of 50 participants had enrolled at time of termination.
Sponsor: Mead Johnson Nutrition (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 6011
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Concentration; Learning

ARMS (2):
- Group 1 - Control A (Experimental): Nutritional beverage containing varying types and levels of carbohydrates
  Interventions: Other: Nutritional Beverage
- Group 2 - Experimental A (Experimental): Nutritional Beverage with varying types and levels of carbohydrates
  Interventions: Other: Nutritional Beverage

INTERVENTIONS:
Other: Nutritional Beverage — Nutritional Beverage with varying types and levels of carbohydrates
  Arms: Group 1 - Control A
Other: Nutritional Beverage — Nutritional beverage with varying types and levels of carbohydrates
  Arms: Group 2 - Experimental A

SUMMARY:
This clinical trial will determine the effect of varying types of carbohydrates on children's concentration.

ELIGIBILITY:
Inclusion Criteria:

* Children 33 months - 39 months

Ages: 33 Months to 39 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Concentration
  Children's ability to concentrate

SECONDARY OUTCOMES:
Attention
  Measures of Attention and Distractibility
Short-Term Memory
  Sentence Repetition
Rule Learning
  Rule Learning Tasks

CONTACTS AND LOCATIONS:
Locations (1):
- Early Cognition Laboratory, Overland Park, Kansas, United States